CLINICAL TRIAL: NCT05036928
Title: Study of MDW Levels Predicting the Development of Sepsis in Hospitalized HIV-infected Patients and Correlation With Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Jun Chen, MD, Deputy Director of Department of Infectious Diseases and Immunology, Shanghai Public Health Clinical Center
Other Study IDs: HIV-MDW
Record Dates: First submitted 2021-09-03; First posted 2021-09-08 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: HIV Infections; Sepsis
MeSH Terms: conditions — HIV Infections; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV infection group
  Interventions: Diagnostic Test: Monocyte distribution width (MDW）

INTERVENTIONS:
Diagnostic Test: Monocyte distribution width (MDW） — All enrolled patients will receive test with MDW.

SUMMARY:
Sepsis is a common and critical complication in HIV-infected patients and an important marker of high risk of patient death. The widely used diagnostic criteria for sepsis still have many deficiencies and do not allow for good prediction and timely determination of the onset of sepsis. In HIV-infected patients, abnormal activation of monocyte-macrophage is also a key mechanism in the development of their sepsis. Monocyte distribution width (MDW) is a marker of the degree of peripheral blood monocyte activation and has been recommended abroad for the early diagnosis of adult sepsis patients in emergency departments. However, in China, MDW has not been applied to the clinic yet, and the related studies are almost blank. Therefore, it is worthwhile to analyze the monocyte activation status of HIV-infected patients by MDW assay and thus predict the occurrence of sepsis.

DETAILED DESCRIPTION:
This is a prospective observational study, and investigators intend to collect HIV-infected patients in our hospital within 1 year from the conduct of this study and hospitalized, after informed consent, for inclusion in the study. Investigators will collect clinical data, basic laboratory indicators, and test MDW levels of the patients and follow the patients until discharge or death.

ELIGIBILITY:
Inclusion Criteria:

* Positive ELISA test results for HIV-1 antibodies;
* Hospitalized patients; Voluntarily signing the patient's informed consent and being able to promise to be followed up;
* No plans to move away from the current trial site during the course of the trial.

Exclusion Criteria:

* Western Blot and/or HIV RNA assay confirmed as HIV negative;
* Women who are pregnant or breastfeeding;
* Current drug users;
* Persons with a history of alcohol abuse that cannot be terminated;
* Persons of non-Chinese nationality;
* Other patients who, in the judgment of the investigator, are deemed unsuitable for participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients hospitalized in our hospital within 1 year since this study was conducted.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with sepsis of admission | within 28 days
  Using Sepsis 3.0 as the diagnostic criteria, the sensitivity and specificity of using MDW to diagnose sepsis in HIV-infected patients.
Number of deaths of enrolled patients | within 28 days
  In HIV infection with sepsis, whether higher MDW score is related to poor prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Crouser ED, Parrillo JE, Seymour CW, Angus DC, Bicking K, Esguerra VG, Peck-Palmer OM, Magari RT, Julian MW, Kleven JM, Raj PJ, Procopio G, Careaga D, Tejidor L. Monocyte Distribution Width: A Novel Indicator of Sepsis-2 and Sepsis-3 in High-Risk Emergency Department Patients. Crit Care Med. 2019 Aug;47(8):1018-1025. doi: 10.1097/CCM.0000000000003799. PMID 31107278
- [Background] Crouser ED, Parrillo JE, Martin GS, Huang DT, Hausfater P, Grigorov I, Careaga D, Osborn T, Hasan M, Tejidor L. Monocyte distribution width enhances early sepsis detection in the emergency department beyond SIRS and qSOFA. J Intensive Care. 2020 May 5;8:33. doi: 10.1186/s40560-020-00446-3. eCollection 2020. PMID 32391157
- [Background] Agnello L, Bivona G, Vidali M, Scazzone C, Giglio RV, Iacolino G, Iacona A, Mancuso S, Ciaccio AM, Lo Sasso B, Ciaccio M. Monocyte distribution width (MDW) as a screening tool for sepsis in the Emergency Department. Clin Chem Lab Med. 2020 Oct 25;58(11):1951-1957. doi: 10.1515/cclm-2020-0417. PMID 32598299
- [Background] Moreira J, Paixao A, Oliveira J, Jalo W, Manuel O, Rodrigues R, Oliveira A, Tinoco L, Lima J, Grinsztejn B, Veloso VG, Japiassu AM, Lamas CC. Accuracy of quick sequential organ failure assessment score to predict mortality in hospitalized patients with suspected infection in an HIV/AIDS reference centre in Rio de Janeiro, Brazil. Clin Microbiol Infect. 2019 Jan;25(1):113.e1-113.e3. doi: 10.1016/j.cmi.2018.08.003. Epub 2018 Aug 15. PMID 30118761
- [Derived] Sun J, Shao Y, Jiang R, Qi T, Xun J, Shen Y, Zhang R, Qian L, Wang X, Liu L, Wang Z, Sun J, Tang Y, Song W, Xu S, Yang J, Chen Y, Tang YW, Lu H, Chen J. Monocyte distribution width (MDW) as a reliable diagnostic biomarker for sepsis in patients with HIV. Emerg Microbes Infect. 2025 Dec;14(1):2479634. doi: 10.1080/22221751.2025.2479634. Epub 2025 Mar 26. PMID 40094401